CLINICAL TRIAL: NCT01453179
Title: Long-term Effects of Aldara® 5% Cream and Solaraze® 3% Gel in the Treatment of Actinic Keratoses on the Face or Scalp With Respect to the Risk of Progression to In-situ and Invasive Squamous Cell Carcinoma
Brief Title: Long-term Effects of Imiquimod and Diclofenac in Actinic Keratoses (LEIDA 2)
Acronym: LEIDA 2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MEDA Pharma GmbH & Co. KG (Industry)
Collaborators: Siro Clinpharm Germany GmbH (until June 2013) (Unknown); Accovion GmbH (Industry)
Responsible Party: Sponsor
Organization: Viatris Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: X-03016-3284; 2010-022054-16 (EudraCT Number)
Record Dates: First submitted 2011-09-30; First posted 2011-10-17 (Estimated); Last update posted 2022-02-07 (Actual); Status verified 2015-04

CONDITIONS: Actinic Keratosis
Keywords: actinic keratosis; invasive SCC; in situ SCC; histological classification; histological progression; clinical clearance; cryotherapy
MeSH Terms: conditions — Keratosis, Actinic | interventions — Imiquimod; Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Aldara 5% Cream (Experimental)
  Interventions: Drug: Imiquimod
- Solaraze 3% Gel (Active Comparator)
  Interventions: Drug: Diclofenac

INTERVENTIONS:
Drug: Imiquimod — One course of treatment (COT) consisting of an overnight application of IMIQ (1 sachet for up to 50 cm2), applied 3 nights per week (e.g. Monday, Wednesday, Friday) for 4 weeks followed by a 4 weeks treatment pause. If necessary, this may be followed by a second COT.
  Arms: Aldara 5% Cream
Drug: Diclofenac — Solaraze® is applied locally to the skin 2 times daily and smoothed into the skin gently. The amount needed depends on the size of the lesion. Normally 0.5 grams (the size of a pea) of the gel is used on a 25 cm2 lesion site. The duration of therapy is 12 weeks.
  Arms: Solaraze 3% Gel

SUMMARY:
This clinical trial serves the purpose to compare the long-term effects of a treatment of actinic keratosis - your skin disorder - using Aldara® 5% cream (Imiquimod) or Solaraze® 3% gel (Diclofenac) on the face or the scalp. In particular, it should be found out whether the healing effect of these two medications on the skin lesions (i.e. the damaged skin parts) can be maintained for a prolonged period.

ELIGIBILITY:
Inclusion Criteria:

To be eligible, a patient must comply with all of the following criteria:

* Immunocompetent patient.
* A study treatment area must be identifiable: Minimum of 5 and maximum of 10 typical visible AKs in one contiguous area of up to 50 cm2 on the face or scalp. The eyelids, the inside of the nostrils or ears, or the lip area inside the vermilion border must not be part of this area.
* A positive histological finding for AK grade I or II. This will be determined from the most suspicious lesion in the STA and there from the most pathological area biopsied during screening visit. This analysis will be done by the central histopathological laboratory.
* Willingness to comply with the obligations of the study.

Exclusion Criteria:

A patient is ineligible and must not enter the study if any of the following criteria is met:

Safety concerns:

* History of hypersensitivity to imiquimod, diclofenac, acetyl salicylic acid, other non steroidal anti-inflammatory drugs (NSAID), hyaluronic acid, or relevant excipients.
* Pregnancy, breast-feeding or planned pregnancy during the study. Women of child bearing potential not using a highly effective method of birth control defined as those which result in a low failure rate (i.e. <1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, hormonal IUDs, tubal ligation or vasectomised partner.

Lack of suitability for the study:

* Presence of AK lesions in the STA with clinically excessive hyperkeratosis as seen in cutaneous horns.
* Any topical AK treatment including imiquimod or diclofenac, or any systemic AK treatment such as systemic retinoids, or any surgical AK treatment at the STA within the last 2 months prior to randomisation.
* Persisting AK lesion at screening visit following topical treatment with imiquimod or diclofenac in the STA.
* Presence of any histologically confirmed skin tumour in the STA: in situ SCC including Bowen's disease, invasive SCC, basal cell carcinoma, or other malignant tumours.
* Any dermatological disease or condition that may exacerbate by treatment with imiquimod or diclofenac (e.g. rosacea, psoriasis, atopic dermatitis).
* Any dermatological disease or condition in the STA that causes difficulty with examination (e.g. eczema).
* Systemic immunomodulatory treatment such as interferon, azathioprine, cyclosporine, retinoids, any oral or injectable corticosteroids, or inhaled or nasal corticosteroids with dosages of >1200 µg/day beclomethasone or equivalent within 4 weeks before start of study treatment.
* History of any malignant tumour with high tumour burden or any systemic antitumour treatment (incl. radiotherapy).
* History of any malignant skin tumour having metastasised or in which metastasis within the study period is likely.
* History of severe cardiovascular, pulmonary, hepatic, renal, gastrointestinal, haematological, endocrine, metabolic, mental, neurological, or other disease within the last two years which might hinder regular treatment and supervision and might lead to premature withdrawal from the study.
* Mentally incapacitated patient.
* Present or history of drug or alcohol abuse within the last 3 years.

Administrative reasons:

* Exposure to an investigational product within the last 3 months.
* Lack of ability or willingness to give informed consent.
* Age below 18 years.
* Lack of willingness to have personal study related data collected, archived or transmitted according to protocol.
* Anticipated non-availability for study visits/procedures.
* Vulnerable subjects (such as persons kept in detention).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2011-10; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Long-term outcome with respect to the risk of progression to SCC (in situ and/or invasive) of treatment with Aldara® 5% cream (IMIQ) and Solaraze® 3% gel (DIC) with increased precision (meta-analysis with study 3271). | 3 years

SECONDARY OUTCOMES:
Recurrence rate | 3 years
Time to recurrence | 3 years
Need of rescue treatment | 3 year
Cosmetic outcome | 3 years
  Cosmetic outcome assessed by patient and investigator on a verbal rating scale.

CONTACTS AND LOCATIONS:
Overall Officials: Ursula Petzold, Dr., Study Director — MEDA Pharma GmbH & Co. KG; Harald Gollnick, Prof. Dr., Principal Investigator — Otto-von-Guericke-University of Magdeburg
Locations (17):
- Austria (3):
  - Medical University Graz, University Clinic for Dermatology and Venerology Graz, Graz
  - Medical Practice, Maria Enzersdorf
  - Medical University Vienna, Department for General Dermatology, Vienna
- Germany (14):
  - Medical Supply Center, Augsburg
  - Licca Clinical Research Institute, Clinic for Dermatolgy and Surgery, Augsburg
  - Medical Practice, Berlin
  - Medical Practice, Dülmen
  - Medical Practice, Germering
  - Medical Department of Otto-von-Guericke-University Magdeburg, University Clinic for Dermatology and Venerology, Magdeburg
  - Medical Practice, Mahlow
  - Department of Dermatology Johannes Gutenberg-University Mainz, Clinical Research Center, Mainz
  - Medical Practice, Markkleeberg
  - Medical Practice for Dermatology and Medical Cosmetics, Mönchengladbach
  - Medical Practice, Münster
  - Derma Center Vechta, Clinic for Dermatology, Vechta
  - Centrovital, Medical Practice for Dermatology, Witten
  - Medical Practice for Dermatology and Venerology, Wuppertal

REFERENCES:
- [Derived] Gollnick H, Dirschka T, Ostendorf R, Kerl H, Kunstfeld R. Long-term clinical outcomes of imiquimod 5% cream vs. diclofenac 3% gel for actinic keratosis on the face or scalp: a pooled analysis of two randomized controlled trials. J Eur Acad Dermatol Venereol. 2020 Jan;34(1):82-89. doi: 10.1111/jdv.15868. Epub 2019 Sep 12. PMID 31407414